CLINICAL TRIAL: NCT05865145
Title: Effects of Two Different Intensities of Aerobic Exercise on Basic Metabolic Panel Perceived Exertion and Exercise Adherence in Older Obese Adults
Brief Title: Effects of Aerobic Exercise on Basic Metabolic Panel Perceived Exertion and Exercise Adherence in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rana Elbanna (Other)
Responsible Party: Sponsor-Investigator, Rana Elbanna, lecturer at faculty of physical therapy at Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR Rana
Record Dates: First submitted 2023-04-05; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Obese; Elderly
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): will receive High Intensity Interval Training program
  Interventions: Device: Electronic Bicycle Ergometer
- Group B (Experimental): will receive Low Intensity Interval Training program
  Interventions: Device: Electronic Bicycle Ergometer

INTERVENTIONS:
Device: Electronic Bicycle Ergometer — Electronic Bicycle equipped with electronic break, display screen, adjustable seat, handle bar and foot straps will be adjusted for High or Low interval intensity training.

SUMMARY:
Participants were randomly assigned to two groups prior to their second visit:

the High intensity interval training group A (HIIT) and Low intensity interval training group B (LIIT).

The randomization processes were conducted in Excel utilizing a random-number generator. Prior to the second visit, each participants' target exercise heart rate ranges were determined.

Group A will receive a program of high intensity interval training program Group B will receive a program of Low intensity interval training program

ELIGIBILITY:
Inclusion Criteria:

* could stand and walk for 30m without becoming out of breath.
* could walk safely without the aid of another person.
* body mass index (BMI) ≥ 30 kg/m2

Exclusion Criteria:

* uncontrolled preexisting health conditions such as:
* uncontrolled hypertension
* uncontrolled diabetes
* uncontrolled heart disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Perceived Exertion | 4 weeks
  The Modified Borg Dyspnea Scale was used to assess perceived exertion during breathing. It was given after the first and final training sessions. The participants were asked to score their difficulty in breathing on a scale of 0 to 10, with 0 indicating no trouble in breathing at all and 10 indicating maximum difficulty in breathing
Exercise Adherence | 4 weeks
  The Exercise Adherence Rating Scale (EARS) is a self-reported 16-item questionnaire that rates adherence to prescribed workouts. The EARS are divided into three components. The suggested exercise questionnaire is discussed in Section (A), Section (B) discusses exercise adherence behavior, and Section (C) discusses the factors for exercise adherence/non-adherence. All items in sections B and C are rated on a 5-point Likert scale (0 = fully agree to 4 = entirely disagree). Section 'B' favourably phrased items (items 1, 4, and 6) and Section 'C' positively phrased items (items 4, 5, 6, and 7) are assessed in reverse order. Sections "B" and "C" have possible total scores ranging from 0 to 24 and 0 to 40, respectively. The potential total score for parts (B) and (C) is 64. A higher total score suggests more adherence to exercise.
Glucose level | 4 weeks
  blood test that examines Glucose level in (mmol/L)
calcium level | 4 weeks
  blood test that examines calcium level in (mg/dL)
sodium level | 4 weeks
  blood test that examines sodium level in (mmol/L)
potassium level | 4 weeks
  blood test that examines potassium level in (millimol/L)
carbon dioxide level | 4 weeks
  blood test that examines carbon dioxide level in parts per million (ppm)
chloride level | 4 weeks
  blood test that examines chloride level in mmol/L
blood urea nitrogen (BUN) level | 4 weeks
  blood test that examines blood urea nitrogen (BUN) level in (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic faculty of physical therapy at Cairo University, Giza, Egypt